CLINICAL TRIAL: NCT05952063
Title: Validation of the Korean Version of Schema Scale of Mental Health Service, MINDLiNG
Brief Title: Validation of Schema Scale of Mental Health Service
Status: Completed | Type: Observational
Sponsor: 40FY (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUH_Schema_Scale
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Mental Health Services; Personality
Keywords: maladaptive schema; mental health problem; personality test; digital mental health service

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Digital Psychological Test: Schema Scale — Thirty-five questionnaire, 5-point likert scale

SUMMARY:
Digital Mental Health Service, MINDLiNG, has developed Schema Scale that identifies individual's personality based on schema theory. The goal of this study is to determine the reliability and validity of the Schema Scale.

DETAILED DESCRIPTION:
Most of the mental health service programs are limited to targeting specific psychiatric symptoms, which does not necessarily consider the personality and characteristics of individuals. To provide more personalized mental health care service, it is essential to identify the personality of individuals through valid psychological test.

Thus, MINDLiNG has developed the Schema Scale based on schema theory and psychodynamic theory in order to provide personalized and evidence-based treatment at the level of psychotherapy.

This study was conducted to evaluate the validity and reliability of the Schema Scale. The scale was administered online on non-clinical population (n = 234). The internal consistency of Schema Scale was evaluated. In addition, its factor structured was studied by exploratory and confirmatory factor analyses. Concurrent validity was examined by comparing the extracted Schema Scale factors with other psychological tests using Pearson's correlation tests.

ELIGIBILITY:
Inclusion Criteria:

* An adult who is able to independently read in Korean and fill out a survey form.

Exclusion Criteria:

* In cases where there is difficulty understanding and reading Korean.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All adults who are willing to complete the online questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Schema Scale | Baseline
  A 35-item questionnaire developed by 40FY for identifying 5-types of maladaptive schema types. The questionnaire consists of 5-point Likert scale. The Schema Scale was developed based on schema theory and other psychodynamic theories. The scale was developed by a certified psychiatrist and 3 clinical psychologists. A higher score for each factor means that the individual has more severe maladaptive psychological schemas.
Perceived Stress Scale (PSS) | Baseline
  The PSS is a 10-item scale that measures the perceived stress on a 5-point severity with higher scores indicating more severe perceived stress.
Self-Efficacy Stress (SES) | Baseline
  The SES is a 23-item scale that assesses the individuals self-efficacy on a 5-point likert scale. Higher scores indicate higher level of self-efficacy.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline
  The CES-D is a 20-item questionnaire that measures depressive symptoms on a 4-point likert scale.
State-Trait Anxiety Inventory (STAI) | Baseline
  The STAI is a 40-item inventory that measures state and trait anxiety. Higher score means higher anxiety.
UCLA Loneliness Scale (UCLA-LS) | Baseline
  A 20-item scale to measure subjective feelings of loneliness as well as feelings of social isolation on a 4-point likert scale.
Short form of the Korean Inventory of Interpersonal Problems Circumplex Scale (KIIP-SC) | Baseline
  A 40-item scale to assess interpersonal problems on a 5-point likert scale.
Diagnostic Test for Personality Disorders - Dependent subscale (DTPD-D) | Baseline
  A 15-item scale to assess dependent personality disorder traits on a 4-point likert scale.
Strait-Trait Anger Expression Inventory (STAXI) | Baseline
  The STAXI is a psychometric assessment that measures state anger, trait anger, and anger expression by 44 items on a 4-point likert scale.
UPPS-P Impulsive Behavior Scale | Baseline
  The scale is composed of 59 items on a 4-point likert scale assessing five factors of impulsivity including negative urgency, lack of premeditation, lack of perseverance, sensation seeking, and positive urgency.
Hewitt Multidimensional Perfectionism Scale (HMPS) | Baseline
  The HMPS is a 45-item measure with three trait subscales measuring self-oriented perfectionism, other-oriented perfectionism, and socially prescribed perfectionism.
State Self-Esteem Scale (SSES) | Baseline
  A 20-item scale on a 5-point likert scale assessing 3 facets of self-esteem: appearance, performance, and social.
Rejection Sensitivity Questionnaire (RSQ) | Baseline
  The RSQ assesses anxious expectations regarding rejection with 18 hypothetical social situations on a 6-point likert scale.
Beck Anxiety Inventory (BAI) | Baseline
  A 21-item self-inventory on a 4-point likert scale measuring common somatic and cognitive symptoms of anxiety.
Intolerance of Uncertainty Scale-Short Form (IUS-12) | Baseline
  A 12-item questionnaire measures responses to uncertain and ambiguous situations that participants rate on a 5-point scale.
Penn State Worry Questionnaire (PSWQ) | Baseline
  The PSWQ is a 16-item self-report questionnaire on a 5-point likert scale designed to measure the trait of worry in adults

CONTACTS AND LOCATIONS:
Overall Officials: Min-Sup Shin, PhD, Principal Investigator — Seoul National University College of Medicine, Department of Psychiatry
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Jeong S, Hwang I, Sung K, Moon W, Shin MS. Validation of a Brief Internet-Based Self-Report Measure of Maladaptive Personality and Interpersonal Schema: Confirmatory Factor Analysis. Interact J Med Res. 2023 Sep 29;12:e48425. doi: 10.2196/48425. PMID 37773606